CLINICAL TRIAL: NCT00390273
Title: Effect of Metformin on Lactate Metabolism in Healthy Subjects
Brief Title: Effect of Metformin on Lactate Metabolism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CRNHRA-06-001; EUDRACT 2006-001348-30
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Hyperlactatemia
Keywords: diabetes; metformin; hyperlactatemia
MeSH Terms: conditions — Hyperlactatemia; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Metformin

SUMMARY:
The main objective of this study is to evaluate the influence of metformin on lactate metabolism.

The main outcome is the lactate production following an exogenous lactate overload in healthy male subjects without metformin and one week later with metformin.

DETAILED DESCRIPTION:
Study design: Physiological study, controlled, open, non randomised

Healthy male subjects, 18 to 30 years old

Principal objective : To evaluate the influence of metformin on lactate metabolism (production) following exogenous lactate overload.

* Objective 2: To evaluate the influence of metformin on lactate metabolism (production) after muscular exercise.
* Objective 3: To evaluate the influence of metformin on lactate metabolism (elimination) after exogenous lactate overload.
* Objective 4: To evaluate the influence of metformin on lactate metabolism (elimination) after muscular exercise.

Principal outcome : Lactate production following exogenous lactate overload.

* Outcome 2: Production of lactate following muscular exercise test.
* Outcome 3 and 3': Parameters modelizing elimination of lactate following exogenous lactate overload (bi-exponential model).
* Outcome 4 and 4': Parameters modelizing elimination of lactate following muscular exercise test (bi-exponential model).

Inclusion criteria:

* Healthy male subjects, 18 to 30 years
* Body mass index (BMI) between 21 and 25 kg/m2 inclusive
* Informed consent

Exclusion criteria :

* Ward of court or under guardianship (sheltered adults)
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalised without their consent
* Person under legal protection
* Existence of a previously diagnosed pathology
* Existence of a metabolic condition (obesity, diabetes) or a family history of such
* Ongoing medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 30 years
* Body mass index (BMI) between 21 and 25 kg/m2 inclusive
* Informed consent

Exclusion Criteria:

* Ward of court or under guardianship (sheltered adults)
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalised without their consent
* Person under legal protection
* Existence of a previously diagnosed pathology
* Existence of a metabolic condition (obesity, diabetes) or a family history of such
* Ongoing medical treatment

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Lactate production following exogenous lactate overload

SECONDARY OUTCOMES:
Production of lactate following muscular exercise test.
Parameters modelizing elimination of lactate following exogenous lactate overload (bi-exponential model).
Parameters modelizing elimination of lactate following muscular exercise test (bi-exponential model).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fontaine, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Centre Hospitalier Universitaire de Grenoble, Grenoble, France